CLINICAL TRIAL: NCT01787253
Title: Microbe-Gut Interaction in Microscopic Colitis and Post-Infectious Irritable Bowel Syndrome (IBS)
Status: Completed | Type: Observational
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Robert Brummer, Dean, Örebro University, Sweden
Other Study IDs: 2010-05; 2010/261 (Other: 2010/261 Uppsala etiknämnd)
Record Dates: First submitted 2010-11-15; First posted 2013-02-08 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Irritable Bowel Syndrome (IBS)
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsies and blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Irritable bowel syndrome (IBS)
- Healthy controls
- Microscopic Colitis (MC)
- Irritable bowel disease (IBD)

SUMMARY:
Objective: This study aims elucidate the pathophysiological link between the environment in the colon (mainly the microbiota), the local immune system and activation of the enteric nervous system in patients with post-infectious IBS (PI-IBS) and microscopic colitis (MC) with special emphasis on microbial-mucosa interactions and evaluation of the effect on the immune activation/response as well as how afferent gut-brain signalling leads to abdominal discomfort.

Method: The project is based on data from three cohorts of patients, one with PI-IBS and one with MC as well as a gender- and age-matched cohort of healthy individuals. Measurement of perceived sensitivity in the gut will be evaluated by pain-response under mechanical stress using a barostat. The HIT (Human intestinal Tissue)-Chip array will be used to characterize the diversity, stability and functionality of the intestinal microbiota on mucosa level, giving a clue to the interactions with the host and insight to changes leading to the development of the two diseases.

Immunohistochemistry and flowcytometry will be used to analyse the location, frequency and phenotype characteristics of lymphoid- and mast cells. Functional analysis of mucosal lymphocytes activated in vitro by products from the intestinal microbiota will be examined by cytokine production using the LuminexTM system. The Ussing chamber technique will allow investigation of the impact of the microbiota and its metabolites on intestinal barrier functions. In this method the sample has access to stressors under standard conditions.

DETAILED DESCRIPTION:
We will make a characterization of lymphocytes, mast cells and gut microflora. Depending on these results we will make stimulations of patient biopsies to find if tissue from patients react differently then patients from healthy.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Healthy and not eating any prescription medication except birth control in pill form

Exclusion Criteria:

* Have or had a history of gastrointestinal disease that has required specialist medical care
* Being lactose intolerance
* Have high blood pressure requiring treatment
* Have premenstrual syndrome
* Lose Weight
* Being pregnant or breast-feed

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from clinic (endoskopimotagningen) at Örebro University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Lymphocyte characterization | After one year of initial infection before treatment
  LPLs and IELs stained with the following flourochrome-conjugated antibodies: anti-CD3-FITC (clone-HIT3a), anti-CD4-FITC/PECy5 (clone-RPA-T4), anti-CD45RA-PE (clone-HI 100), anti-CD45RO-PECy5 (clone-UCHL1), anti-CD19-PE (clone-HIB19) and anti-CD138-FITC (clone-MI15), all from BD Pharmingen (San Diego, CA, USA). Anti-CD8α-ECD (clone-SFCI21Thy2D3) and anti-CD8β-PECy5 (clone-2ST8.5 H7) were purchased from Beckman Coulter (Fullerton, CA, USA) whereas anti-CD38-PECy5 (clone-HIT2), anti-αβTCR-PECy5 (clone-IP26) and anti-γδTCR-PE (clone-B1) were purchased from Biolegend (San Diego, CA, USA). Fluorochrome-conjugated isotype matched control antibodies were used as controls for non-specific staining, and were purchased from BD Pharmingen or Beckman Coulter (IgGκ-FITC, IgG2bκ-PE, IgG1-ECD, IgG2bκ-PECy5, IgG2κ-FITC, IgG1κ-PE, IgG1κ-PECy5, and IgG2a-PECy5).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Brummer, MD, PhD, Principal Investigator — Örebro Universitet
Locations (1):
- Örebro University Hospital, Örebro, Närke, Sweden